CLINICAL TRIAL: NCT04352439
Title: Aspirin for Prevention of Venous Thromboembolism Among Ovarian Cancer Patients Receiving Neoadjuvant Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00105081
Record Dates: First submitted 2020-04-13; First posted 2020-04-20 (Actual); Results first posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Venous Thromboembolism; Ovarian Cancer
MeSH Terms: conditions — Venous Thromboembolism; Ovarian Neoplasms | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aspirin (Experimental): Patients with a Khorana risk score of 1 receive 81 mg aspirin daily while receiving neoadjuvant chemotherapy for ovarian cancer.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — 81 mg aspirin daily

SUMMARY:
This is a pilot study to determine the safety and efficacy of low dose aspirin for the prevention of venous thromboembolism among women with advanced ovarian cancer receiving neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Subjects who are receiving neoadjuvant chemotherapy for advanced epithelial ovarian cancer, including primaries of mullerian, peritoneal, or fallopian tube origin, with a Khorana score of 1 will be recruited from the Duke Gynecology Oncology clinic at Duke Cancer Institute. After discussion of the risks and benefits, written informed consent will be obtained for initiation of prophylactic, daily low dose aspirin (81 mg) therapy. Subjects will receive aspirin tablets in medication vials obtained from the Duke pharmacy supply and will be instructed to take one tablet daily until the day of their interval debulking surgery. The primary outcomes will be safety and medication adherence. Secondary outcome will be rate of VTE. We hypothesize that daily low dose aspirin will be safe with acceptable medication adherence and may reduce the incidence of venous thromboembolic events during neoadjuvant chemotherapy for low risk patients when compared to a historical control.

Adverse safety events and medication adherence will be evaluated using descriptive statistics using a validated questionnaire. We will calculate the incidence of venous thromboembolism among the study cohort and estimate a 95% exact binomial confidence interval. A drop greater than 20% (from 8% in the historical control to 6.4%) in the venous thromboembolism rate would be considered clinically meaningful. We will also monitor for adverse safety events related to low dose aspirin use, including major or minor bleeding events, clinically significant thrombocytopenia (resulting in treatment delay), and gastrointestinal complications. Of note, low dose aspirin for venous thromboembolism prevention is already considered an acceptable option for standard of care for patients with multiple myeloma receiving antiangiogenesis agents with chemotherapy and/or dexamethasone as well as for postoperative thromboprophylaxis for some orthopedic procedures; we therefore believe the potential benefit outweighs any clinically significant risks.

Subjects will be recruited from patients at the Duke Gynecology Oncology clinics at the Duke Cancer Center or Macon Pond (Duke Women's Cancer Care Raleigh) with advanced epithelial ovarian cancer, including primaries of mullerian, peritoneal, or fallopian tube origin, who are going to initiate neoadjuvant chemotherapy. A provider will approach the patient and inquire about interest in participating in the study. If the patient desires to receive more information about participating, clinical research personnel will discuss the study with patient and obtain informed consent if all selection criteria are met (detailed in a prior section). If the patient consents, they will then be considered an enrolled study subject. We will use the Duke hosted REDCap platform for collecting eConsent. If the patient is willing to hear about the study but a member of the research team is unable to be physically present in clinic, the research team will contact the patient via phone to perform the same recruitment, eligibility screening, and consent process that would typically be completed in person.

An estimated 120 patients will receive neoadjuvant chemotherapy for advanced ovarian cancer at Duke Gynecology Oncology clinics for the designated study recruitment period of 07/01/2020 to 12/30/2021 with an estimated 50% accrual rate for a total of 60 enrolled patients. Currently there is no established practice guideline for venous thromboembolism prophylaxis for these high risk patients. There will be no direct cost to subjects for participation in the study. They will not incur any costs for travel as they will already be presenting to Duke Gynecology Oncology clinic for their scheduled clinic visit. The study drug will be provided without cost. There will be additional time (10 minutes) incurred with study participation for informed consent and explanation of the study design and medication adherence diary. Subjects will not be compensated.

ELIGIBILITY:
Inclusion Criteria:

* Khorana score = 1
* Over age 18
* English-speaking female patients
* Able to consent
* Receiving neoadjuvant chemotherapy Cancer of primary ovarian, fallopian tube, mullerian, or peritoneal origin

Exclusion Criteria:

* Allergy or intolerance to study medication
* Indication for a non-aspirin form of antiplatelet (i.e. cardiac stent)
* Already on alternative form of anticoagulation
* Active bleeding
* High risk for active bleeding (i.e. recent intracranial bleed or gastrointestinal bleed, known brain metastases)
* Thrombocytopenia (platelets <50,000)
* Unable to complete medication adherence diary
* Unable to take oral medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-08-08 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Davidson, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Sarasota Memorial HealthCare System, Sarasota, Florida
  - Duke University Hospital, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salinaro JR, McQuillen K, Stemple M, Boccaccio R, Ehrisman J, Lorenzo AM, Havrilesky L, Secord AA, Galvan Turner V, Moore KN, Davidson B. Incidence of venous thromboembolism among patients receiving neoadjuvant chemotherapy for advanced epithelial ovarian cancer. Int J Gynecol Cancer. 2020 Apr;30(4):491-497. doi: 10.1136/ijgc-2019-000980. Epub 2020 Feb 12. PMID 32054646
- [Background] Faour M, Piuzzi NS, Brigati DP, Klika AK, Mont MA, Barsoum WK, Higuera CA. Low-Dose Aspirin Is Safe and Effective for Venous Thromboembolism Prophylaxis Following Total Knee Arthroplasty. J Arthroplasty. 2018 Jul;33(7S):S131-S135. doi: 10.1016/j.arth.2018.03.001. Epub 2018 Mar 8. PMID 29656974
- [Background] Key NS, Khorana AA, Kuderer NM, Bohlke K, Lee AYY, Arcelus JI, Wong SL, Balaban EP, Flowers CR, Francis CW, Gates LE, Kakkar AK, Levine MN, Liebman HA, Tempero MA, Lyman GH, Falanga A. Venous Thromboembolism Prophylaxis and Treatment in Patients With Cancer: ASCO Clinical Practice Guideline Update. J Clin Oncol. 2020 Feb 10;38(5):496-520. doi: 10.1200/JCO.19.01461. Epub 2019 Aug 5. PMID 31381464

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aspirin
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aspirin
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Venous Thromboembolism
Time Frame: Up to six months
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin
Number analyzed (Participants) | 19
Participants | 4

2. Primary Outcome: Number of Participants With at Least One Adverse Event
Description: Adverse events will only include those that are determined to be related to the study drug.
Time Frame: Up to six months
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin
Number analyzed (Participants) | 19
Participants | 0

3. Primary Outcome: Medication Adherence
Description: Patient adherence to aspirin as defined by percent of pills used.
Time Frame: Up to six months
Population: Data not collected.
Arm/Group | Aspirin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months with an average of 2.5 months.
Description: Patient records were reviewed regularly for adverse events.
Arm/Group | Aspirin
All-Cause Mortality (participants affected / at risk) | 8/19
Serious Adverse Events (participants affected / at risk) | 6/19
Other Adverse Events (participants affected / at risk) | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=19)
DVT (Vascular disorders) | 4 (4)
sepsis (Blood and lymphatic system disorders) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT04352439/Prot_SAP_002.pdf
  • Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT04352439/ICF_001.pdf